CLINICAL TRIAL: NCT01613937
Title: Dulce Mothers: A Community Approach to Reduce the Risks of Developing Diabetes After Gestational Diabetes
Brief Title: Community Approach to Reduce the Risks of Diabetes After Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Primary Investigator, Scripps Whittier Diabetes Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SWDI Dulce Mothers
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes
Keywords: Latinas; Gestational Diabetes; Prevention
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle (Experimental): 12 once weekly Lifestyle training program
  Interventions: Behavioral: Dulce Mother lifestyle training program

INTERVENTIONS:
Behavioral: Dulce Mother lifestyle training program — 12 once weekly culturally tailored lifestyle management sessions

SUMMARY:
Objective: The current study examined the effectiveness of a culturally-appropriate adaptation of the diabetes prevention program (DPP) curriculum in reducing type 2 diabetes risk in Latinas with a history of gestational diabetes mellitus (GDM).

Research Design and Methods: Seventy-six Latinas aged 18-45 years with GDM in the past 3 years participated in an 8-week group-based, peer-educator led lifestyle intervention based on the DPP, with adaptations appropriate to Latino culture and recent mothers. Clinical and self-report indicators were assessed at baseline, post-intervention (month-3), and follow-up (month-6).

Hypothesis-The modified culturally tailored DPP will improve risk factors associated with the development of type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Latina
* GDM within the last 3 years
* able and willing to participate in physical activity sessions

Exclusion Criteria:

* current diabetes
* severe illness that would preclude them from coming to the sessions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months

SECONDARY OUTCOMES:
weight | 6 months
lipids | 6 months
blood pressure | 6 months
composition of dietary intake at all time points | 6 months
hours of physical activity per week at all time points | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute